CLINICAL TRIAL: NCT05876403
Title: Effects of Respiratory Proprioceptive Neuromuscular Facilitation (PNF) Technique on Pulmonary Function of Chronic Pulmonary Obstructive Disease (COPD) Patients.
Brief Title: Respiratory Proprioceptive Neuromuscular Facilitation Technique in Chronic Pulmonary Obstructive Disease Patients.
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Maira Tamkeen
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: COPD
Keywords: Peak Expiratory Flow Rate (PEFR); Pulmonary function; PNF techniques
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): The protocol for controlled group will consist of 35-60years old participants with moderate to severe COPD.
  At baseline measurements will be collected and COPD assessment test (CAT) and Modified Borg Scale will be taken. Participants will then be made to perform breathing and aerobic exercises (3sessions per week) for 6 weeks and after every 2 weeks outcome measures will be evaluated using chest expansion, spirometry, and 6 minutes walk test (6MWT) along with CAT and Modified Borg Scale.
  Interventions: Other: Conventional
- PNF Techniques (Experimental): The same protocol will be followed for the 30 participants of experimental group where after the baseline measurements, participants will perform breathing and aerobic exercises along with PNF techniques (3 sessions per week for 6 weeks). The outcome Measures will be measured after every 2 weeks through Spirometry, CAT, Modified Borg Dyspnea Scale and 6 minutes walk test
  Interventions: Other: PNF

INTERVENTIONS:
Other: Conventional — The participants of controlled group will be given the treatment protocol after baseline measurements controlled breathing techniques (3session per week 10mins for 6 weeks) & Aerobic exercise(3 session per week for 6 weeks) with 10sec hold into 10reps.outcome measures will be recorded through a digital spirometer & measurement of 6MWT & chest expansion.
  Arms: Conventional
Other: PNF — The participants of experimental group will be given the Intervention protocol after baseline measurements. Additionally these 30 participants will also receive PNF technique exercises consisting of Thoracic Vertebral pressure, Anterior Basal stretch, and Intercostal stretch for 20-25 minutes in 3 sessions per week, and outcomes Measures will be recorded through a digital spirometer and measurements of 6 minutes walk test and chest Expansion.
  Arms: PNF Techniques

SUMMARY:
The purpose of this study is to evaluate the impact of PNF technique combined with aerobic exercises among COPD patients in a clinical setting. Previous literature has evaluated this technique in ventilated patients but in clinical setting specifically in Pakistan, this invention therapy has not been implied in COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disorder manifested as breathlessness, respiratory difficulties and persistent cough is one of the biggest causes of mortality around the world. 2.1% of Pakistani population has COPD. Proprioceptive neuromuscular facilitation is used as management technique in which muscle stretching promotes chest wall mobility and restores regular breathing rhythm. In previous studies, PNF technique combined with aerobic exercises has been utilized to improve Pulmonary functions in COPD patients. But the sample size of these studies was small and participants were ventilated patients, hence not targeting the diaphragm. Our study shall evaluate the impact of PNF technique combined with aerobic training on the Pulmonary function of COPD patients in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Both male & female participants.
* Diagnosed COPD patients
* Age 35-60years
* Ratio of forced expiratory volume in first second & forced vital capacity(FEV1/FVC <0.7,30%<FEV1<80%
* Stable clinical condition.

Exclusion Criteria:

* Serious conditions with require supplementary oxygen or ventilator/support devices.
* COPD exacerbation within last 4weeks
* Patients with recent chest wall trauma, surgery or deformity.
* Patient with neurological, psychological, musculoskeletal, or cardiac medical history.
* Pulmonary disease with physical impairment.
* Inability to follow the pulmonary rehabilitation program.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | two weeks
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | two weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
  Changes in FVC from baseline to 5th and after 15th day of intervention will be assessed.
Forced expiratory volume in 1sec (FEV1) | two weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal
Chest Expansion | two weeks
  The expansion of chest during breathing will be measures and axillary, nipple and xiphisternal level using a measuring tape.
Modified Borg Dyspnea Scale | two weeks
  Participants will fill this 12 points Scale to show breathing difficulty from 0 to 10.
COPD assessment test | two weeks
  8 points questionnaire will evaluate patients Pulmonary function capacity through semantic 6 point difference Scale.

SECONDARY OUTCOMES:
6 minutes walk test: | two weeks
  This test with minimum important distance of 25 metres will assess aerobic & functional capacity of participants in a 6 minutes walk.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Islamabad, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Putt MT, Watson M, Seale H, Paratz JD. Muscle stretching technique increases vital capacity and range of motion in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2008 Jun;89(6):1103-7. doi: 10.1016/j.apmr.2007.11.033. PMID 18503806
- [Background] Liu K, Yu X, Cui X, Su Y, Sun L, Yang J, Han W. Effects of Proprioceptive Neuromuscular Facilitation Stretching Combined with Aerobic Training on Pulmonary Function in COPD Patients: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2021 Apr 13;16:969-977. doi: 10.2147/COPD.S300569. eCollection 2021. PMID 33880021
- [Background] Reddy RS, Alahmari KA, Silvian PS, Ahmad IA, Kakarparthi VN, Rengaramanujam K. Reliability of Chest Wall Mobility and Its Correlation with Lung Functions in Healthy Nonsmokers, Healthy Smokers, and Patients with COPD. Can Respir J. 2019 Feb 25;2019:5175949. doi: 10.1155/2019/5175949. eCollection 2019. PMID 30931074
- [Background] Make BJ, Yawn BP. Breathing Life Into COPD Management: Ongoing Monitoring, Pulmonary Rehabilitation, and Individualized Care. Chest. 2018 Oct;154(4):980-981. doi: 10.1016/j.chest.2018.08.1023. PMID 30290931